CLINICAL TRIAL: NCT00100191
Title: EMMY Trial: a Randomized Comparison of Uterine Artery Embolization and Hysterectomy for the Treatment of Symptomatic Uterine Fibroids
Brief Title: Emmy Trial: Uterine Artery Embolization (UAE) Versus Hysterectomy for Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Collaborators: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NWO-DO 945-01-17
Record Dates: First submitted 2004-12-23; First posted 2004-12-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-12

CONDITIONS: Menorrhagia; Leiomyoma; Uterine Neoplasms
Keywords: hysterectomy; fibroids; uterine artery embolization; therapeutic embolization; uterus; menorrhagia
MeSH Terms: conditions — Menorrhagia; Leiomyoma; Uterine Neoplasms | interventions — Uterine Artery Embolization; Hysterectomy

INTERVENTIONS:
Procedure: uterine artery embolization
Procedure: hysterectomy

SUMMARY:
The Emmy trial is set up to evaluate the safety and efficacy of uterine artery embolization (UAE) in comparison to hysterectomy for the treatment of symptomatic uterine fibroids. UAE was considered equivalent to hysterectomy when at least 75% of patients had normalization of heavy menstrual blood loss after treatment.

DETAILED DESCRIPTION:
Uterine Artery Embolization (UAE) is a new treatment for heavy menstrual bleeding caused by uterine fibroids. UAE is already being performed on a regular basis, without profound evidence: no good quality randomized controlled trials have been conducted. The EMMY trial evaluates the safety and efficacy of UAE in a randomized comparison to hysterectomy. Patients were included when they had uterine fibroids and menorrhagia, and were eligible for hysterectomy. The primary endpoint is the elimination of menorrhagia after a two-year follow-up period. Secondary endpoints comprise: effect on complaints of pain and pressure, quality of life issues, uterine volume reduction, effect on ovarian function and cost-effectiveness. Patients were randomly assigned to either UAE or hysterectomy (1:1). All patients were followed for two years after treatment. Whether UAE can be an alternative to hysterectomy as treatment of first choice depends on the balance of efficacy, costs, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Uterine fibroids
* Menorrhagia
* Scheduled for hysterectomy
* Pre-menopausal

Exclusion Criteria:

* Childwish (planning to conceive)
* Pregnancy
* Suspected malignancy
* Untreated pelvic inflammatory disease (PID)
* Clotting disorders
* Contrast fluid allergy
* Presence of intrauterine device (IUD)
* Renal failure (creatinine > 150 mmol/l)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-02; Study Completion 2006-04

PRIMARY OUTCOMES:
The primary endpoint is the normalization of menorrhagia after a two-year follow-up period

SECONDARY OUTCOMES:
Effect on complaints of pain and pressure
Technical failure
Complications
Quality of life issues
Uterine volume reduction
Effect on ovarian function
Cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: J.A. Reekers, MD, PhD, Principal Investigator — Academic Medical Centre, Department of Radiology
Locations (2):
- Netherlands (2):
  - Academic Medical Centre Amsterdam, Amsterdam
  - 27 Other Participating Hospitals of Varying Sizes Throughout the Country, Amsterdam

REFERENCES:
- [Result] Hehenkamp WJ, Volkers NA, Van Swijndregt AD, De Blok S, Reekers JA, Ankum WM. Myoma expulsion after uterine artery embolization: complication or cure? Am J Obstet Gynecol. 2004 Nov;191(5):1713-5. doi: 10.1016/j.ajog.2004.02.001. PMID 15547547
- [Derived] Hehenkamp WJ, Volkers NA, Bartholomeus W, de Blok S, Birnie E, Reekers JA, Ankum WM. Sexuality and body image after uterine artery embolization and hysterectomy in the treatment of uterine fibroids: a randomized comparison. Cardiovasc Intervent Radiol. 2007 Sep-Oct;30(5):866-75. doi: 10.1007/s00270-007-9121-7. PMID 17671809
- See also: Information site of the Emmy trial for patients (in Dutch) — http://www.emmystudie.nl